CLINICAL TRIAL: NCT01830270
Title: Preoperative Chemotherapy With Weekly Cisplatin, Epirubicin and Paclitaxel (Intensified PET) in Patients With Locally Gastric Cancer : a Phase II Proof-of-concept Study.
Brief Title: Preoperative Dose-dense Chemotherapy With Weekly Cisplatin, Epirubicin and Paclitaxel to Treat Patients With Locally Gastric Cancer
Acronym: IPEC-GC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPEC-GC
Record Dates: First submitted 2012-03-08; First posted 2013-04-12 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2016-01

CONDITIONS: Stomach Neoplasms; Oesophageal Junction Cancer; Lower Oesophagus Cancer
Keywords: medical oncology; chemotherapy optimization; dose density
MeSH Terms: conditions — Stomach Neoplasms | interventions — Epirubicin; Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET regimen (Experimental)
  Interventions: Drug: Epirubicin; Drug: Cisplatin; Drug: Paclitaxel; Procedure: gastric surgery

INTERVENTIONS:
Drug: Epirubicin — 8 weekly cycles of chemotherapy with epirubicin (50 mg/m2)associated with cisplatin and paclitaxel with a break of one week without chemotherapy between cycle 4 and 5.
Drug: Cisplatin — 8 weekly cycles of chemotherapy with cisplatin (30 mg/m2) associated with epirubicin and paclitaxel with a break of one week without chemotherapy between cycle 4 and 5.
Drug: Paclitaxel — 8 weekly cycles of chemotherapy with paclitaxel (90 mg/m2) associated with epirubicin and paclitaxel with a break of one week without chemotherapy between cycle 4 and 5.
Procedure: gastric surgery — surgery will be scheduled within 4-6 weeks after the end of the last cycle of chemotherapy.

SUMMARY:
If surgery remains the main treatment for gastric cancer without distant metastases; perioperative-chemotherapy increased the likelihood of progression free survival. Perioperative chemotherapy appears to have many advantages : to reduce the tumor volume, to improve the R0 resection rate, and to act on micro-metastases. Therefore, peri-operative chemotherapy combining cisplatin, epirubicin and 5-Fluorouracile is a validated strategy to treat gastric cancer. However, several pitfalls remained. Particularly, only 42% of patients could received post-chemotherapy, due to post-operative complications and toxicities. To overcome this limitation, the investigators will conduct a phase II clinical trial assessing the clinical interest of a dose-dense preoperative chemotherapy combining cisplatin (P), epirubicin (E) and paclitaxel (T). The increasing evidence of taxane's role in gastric cancer treatment, as well as the biological synergisms reported in paclitaxel/cisplatin and paclitaxel/epirubicin combinations, sustain the development of dose density based on PET combination in gastric carcinoma. The aim of the IPEC-GC study is to evaluate the effectiveness of this PET preoperative regimen

DETAILED DESCRIPTION:
The IPEC-GC study is a proof-of-concept study evaluating the efficacy and feasibility of PET regimen in 61 patients with lower oesophagus, oesophagus junction or gastric carcinoma.

Preoperative chemotherapy include eight weekly preoperative cycles of cisplatin (30mg/m2), epirubicin (50 mg/m2) and paclitaxel (90 mg/m2)with a break of one week without chemotherapy between cycle 4 and 5. Surgery is performed within 4-6 weeks after the end of the last cycle of chemotherapy. Primary endpoint of this trial is the curative resection rate (=R0). R0 must be higher than the 79% achieved in previous published studies. Response rate, histologic response rate (Becker score), progression-free survival, overall survival, impact of complete response in survival and dose-density are secondary endpoints. For an ancillary study, tumors (biopsies and operative specimens) and sera will be collected to identify biomarkers correlated with treatment efficacy.

This study is carried out by the Besançon University Hospital and were approved by the independent Est-II ethics committee and by the French National Authority for Health: AFSSAPS.

ELIGIBILITY:
Inclusion criteria :

* Age > 18 and < 70 years (male and female)
* surgical resectability
* ECOG performance status ≤ 1
* ASA score < 3 (appreciation by a surgeon)
* BMI < 30 if an upper oesogastrectomy is required
* no previous cytotoxic chemotherapy
* ejection fraction > 50% in echocardiography before start of therapy
* written informed consent

Non-inclusion criteria :

* distant metastases or infiltration of adjacent structures or organs and all primarily not resectable stages
* relapse
* hypersensitivity against Paclitaxel, Epirubicin or Cisplatin
* malignant secondary disease, dated back < 5 years (exception: in situ carcinoma of the cervix uteri, adequately treated skin basal cell carcinoma)
* peripheral polyneuropathy
* diabetes complicated by coronary artery disease or vasculopathy
* Severe respiratory insufficiency
* patient with weight loss > 10%
* pregnancy or lactation
* inclusion in another trial
* patient with any medical or psychiatric condition or disease which would make the patient inappropriate for entry into this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2015-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
curative resection rate | an expected average of 4 weeks after surgery

SECONDARY OUTCOMES:
response rate | between 2 and 4 weeks after the end of the last cycle of chemotherapy
  Response rate will be evaluated using RECIST v1.1 criteria (Response Evaluation Criteria in Solid Tumors ; Eisenhauer et al, 2009) by a CT-scan done between 2 and 4 weeks after the end of the last cycle to verify the absence of local or distant progression before surgery
histologic response rate | an expected average of 4 weeks after surgery
  Histologic response rate will be determined by the pathologist laboratory on operative specimens using Becker's score (Becker et al, 2003) to measure effects of neoadjuvant chemotherapy on gastric cancer.
tolerance of the therapeutic association | 1 week after each chemotherapy cycle
  Toxicities will be evaluated using Common Terminology Criteria for Adverse Events version 4.
progression free survival | from date to initiation of chemotherapy until the date of first documented progression (within 5 years after surgery)
global survival | from date to initiation of chemotherapy until the date of death for any cause (within 5 years after surgery)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - University hospital of Besançon, Besançon
  - FNLCC center Georges François Leclerc, Dijon
  - Hospital of Belfort-Montbeliard, Montbéliard

REFERENCES:
- [Result] Jary M, Ghiringhelli F, Jacquin M, Fein F, Nguyen T, Cleau D, Nerich V, El Gani M, Mathieu P, Valmary-Degano S, Arnould L, Lassabe C, Lamfichekh N, Fratte S, Paget-Bailly S, Bonnetain F, Borg C, Kim S. Phase II multicentre study of efficacy and feasibility of dose-intensified preoperative weekly cisplatin, epirubicin, and paclitaxel (PET) in resectable gastroesophageal cancer. Cancer Chemother Pharmacol. 2014 Jul;74(1):141-50. doi: 10.1007/s00280-014-2482-0. Epub 2014 May 14. PMID 24824852